CLINICAL TRIAL: NCT01876017
Title: An Open Labeled Clinical Study to Evaluate the Safety and Efficacy of of Bone Marrow Derived Mono Nuclear Stem Cell (BMMNCs) in Chronic Renal Failure Patients. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of BMMNC in Patients With Chronic Renal Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Sub Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BMCRF/2013//01
Record Dates: First submitted 2013-06-08; First posted 2013-06-12 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Renal Failure
Keywords: CRF; STEM CELL; CKD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMMNC (Other): Intravenous transfer of Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)
  Interventions: Biological: Intravenous transfer of Autologous (BMMNCs)

INTERVENTIONS:
Biological: Intravenous transfer of Autologous (BMMNCs) — Intervention therapy , Total 3 doses ,in 30 days ,in 7days interval Intravenous transfer of Autologous (BMMNCs)

SUMMARY:
This Study is single arm, single center trial to check the safety and efficacy of Autologous Bone Marrow derived Mono Nuclear Stem Cell (BMMNCs)for the patient with CRF

DETAILED DESCRIPTION:
Chronic kidney failure, also called chronic kidney disease, describes the gradual loss of kidney function. Kidney failure is a medical condition in which kidneys fail to filter metabolic wastes and toxins out of the body and a series of symptoms will be developed .It is common, frequently un recognised and often exists together with other conditions (for example, cardiovascular disease and diabetes). When advanced, it also carries a higher risk of mortality. The risk of developing CKD(Chronic Kidney diseases ) increases with increasing age, and some conditions that coexist with CKD become more severe as kidney dysfunction advances CKD can progress to established renal failure in a small but significant percentage of people. This classification divides CKD into five stages. Stages 3-5 may be defined by glomerular filtration rate (GFR) alone, whereas stages 1 and 2 also require the presence of persistent proteinuria, albuminuria or haematuria, or structural abnormalities.

Stem cells have two important characteristics that distinguish them from other types of cells. First, they are unspecialized cells that renew themselves for long periods through cell division. The second is that under certain physiologic or experimental conditions, they can be induced to become cells with special function such as the beating cells of heart muscle or the insulin- producing cells of the pancreas as well as the neurons of brain.So our approach is to prove safety and efficacy of stem cell in CRF

ELIGIBILITY:
Inclusion Criteria:

* Age limit: 18 -65
* willingness to undergo Bone marrow and umbilical cord derived Mesenchymal stem cell transplantation.
* To give an informed consent as well as sign the required Informed Consent Form (ICF) for the study.
* willingness to regularly visit the hospital / clinic for follow up during the follow up period / on prior agreed time points as per the protocol.

Exclusion Criteria:

* Patients with pre-existing or current systemic disease such as lung , liver (exception: history of uncomplicated hepatitis A) gastrointestinal , cardiac, immunodeficiency (including HIV) or any other condition determined by history or laboratory investigation that could cause a neurological defect (including syphilis, clinically relevant polyneuropathy) etc.
* Women who are pregnant or lactating
* Chronic kidney disease due to autoimmune aetiology, connective tissue disease, amyloidosis and storage disorders.
* Suffering from Severe co-morbidities like cardiac insufficiency, congestive cardiac failure, malignancy, infection, sepsis and bed sores.
* Positive test results for HIV and AIDS complex ,HCV (hepatitis C virus ), HbsAg and Syphilis
* Hemoglobin level below 7g %
* estimated glomerular filtration rate (eGFR) of < 45ml/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maintain or demonstrate improvement in laboratory values. | 3 month
  • Hematological (Complete blood count (CBC) Complete blood count (CBC) urea(mg/dL), creatinine (mg/dL), plasma calcium(mg/dL), plasma alkaline phosphatase (U/L),plasma phosphorus (mg/dL), plasma cholesterol(mg/dL), plasma HDL-cholesterol (mg/dL), plasma triglyceride (mg/dL), hematocrit (%) and erythrocyte(M/_L) values were evaluated before and at the end of the study.)

SECONDARY OUTCOMES:
pain intensity by VAS | 3 month
  Assessment of pain by visual analogue score
Improvement in SF36(Short form 36) score | 3 month
  The SF36, a short-form QoL scoring system with 36 items, is a self-administered questionnaire that was constructed to fill the gap between much more lengthy surveys and relatively coarse single-item measures of the QoL
Improvement in subjective global assessment | 3 month
the incident of uremia and dialysis requirement | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India